CLINICAL TRIAL: NCT07024719
Title: First Use of Duke 4D Microscope Integrated OCT (MIOCT) Integrated Into Zeiss Artevo 800 Ophthalmic Surgical Microscope in the Operating Room
Brief Title: 4D Duke Microscope Integrated Optical Coherence Tomography in a Zeiss Artevo 800
Acronym: 4D MIOCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00117756
Record Dates: First submitted 2025-05-28; First posted 2025-06-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Corneal Diseases; Retinal Diseases; Ocular Diseases
Keywords: Microscope integrated OCT; intraoperative OCT; optical coherence tomography (OCT)
MeSH Terms: conditions — Corneal Diseases; Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Group 1 - Imaging during ophthalmic surgery (Experimental): Research 4D MIOCT imaging will be performed in the operating room during clinically-indicated surgical procedures. Imaging will be of one or both eyes.
  Interventions: Device: 4D MIOCT integrated into a Zeiss Artevo 800

INTERVENTIONS:
Device: 4D MIOCT integrated into a Zeiss Artevo 800 — 4D MIOCT integrated into a Zeiss Artevo 800 surgical microscope with an add-on investigational 3D OCT scanner

SUMMARY:
The study team will conduct the first in-human pilot studies using 4D MIOCT for imaging in the operating room. Building on the earlier integration and wet-lab validations, the researchers will assess the system's ease of use, safety, and visualization of intended structures during various anterior and posterior segment ophthalmic procedures.

DETAILED DESCRIPTION:
The purpose of this project is to capture research images from microscope integrated Optical Coherence Tomography (MIOCT) integrated into a Zeiss Artevo 800 surgical microscope with an add-on investigational 3D OCT scanner (hereafter called the 4D MIOCT) in participants undergoing clinically-indicated surgical procedures for a range of ocular diseases. The researchers will evaluate normal and abnormal microanatomy of the eye, image during surgical procedures, and track subretinal injections for therapeutic delivery during surgery (volumes measured/analyzed from the OCT images after surgery).

This study is an observational imaging study with no treatment interventions for research purposes. The population is 5 adult ophthalmic surgical patients scheduled for eye surgery at Duke Eye Center, Durham. Up to 8 patients may be enrolled due to potential for surgery scheduling changes that would not allow research imaging on a surgery day for up to 3 patients. Research activities consist of investigational 4D MIOCT integrated into Zeiss Artevo 800 imaging of the eyes during surgery and collection of clinical data and other imaging from the participant's medical record, clinical visit and surgical procedure.

Additional imaging of the participant's eye performed for clinical care will be extracted from the medical record for comparison to the intraoperative images. In this initial pilot, comparisons will enable design of future studies for accuracy, precision and reproducibility of the research device in eye surgery.

For study participants there is no additional risk to the participant beyond what is normal for their ophthalmic surgery. No medications or surgical interventions/activities will be performed for research purposes.

Images will be captured during the standard care ophthalmic microsurgery.

This research will utilize the data gathered during OCT imaging performed as described above. The data collected from the OCT systems will be analyzed offline to allow for image processing and alternate visualizations of the area under study. The data gathered from 4D MIOCT imaging will be compared to existing clinical studies (performed as part of standard of care) on the participant, should they exist, for the purpose of identifying whether new information is gained by 4D MIOCT. Researchers will review the participant's Medical Record for up to three eye care visits prior to surgery and record information related to ocular health, eye examinations and imaging and prior ophthalmic treatment. No additional clinical studies will be performed for the purpose of this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants 18 years of age and older
* Patients undergoing surgery for ocular disease
* Adults able and willing to give informed consent to participate in the study

Exclusion Criteria:

* Patients with any ocular disease that restricts the ability to perform OCT scanning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
4D MIOCT ease of use | Standard of care visit - day 1
  Determining subjective operator comfort and satisfaction using Likert Scales (Likert scores 1-5)

SECONDARY OUTCOMES:
Surgical workflow | Standard of care visit - day 1
  Evaluation of surgical workflow/interference using Likert Scales (Likert scores 1-5)
Presence of microanatomy as measured by 4D MIOCT image reading | Standard of care visit - day 1
  Presence (Yes/No) of retinal anatomy as measured from 4D MIOCT grading
Presence of abnormal microanatomy as measured by 4D MIOCT | Standard of care visit - day 1
  Combination of presence (Yes/No) and severity (e.g. mild, moderate, severe) of abnormal retinal structures and measured from 4D MIOCT images

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Toth, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
This is a first in-human pilot study using 4D MIOCT in the operating room. There will only be 5 participants enrolled in this study. If further studies are performed after this pilot, we may share IPD.

REFERENCES:
- [Background] Carrasco-Zevallos OM, Keller B, Viehland C, Shen L, Seider MI, Izatt JA, Toth CA. Optical Coherence Tomography for Retinal Surgery: Perioperative Analysis to Real-Time Four-Dimensional Image-Guided Surgery. Invest Ophthalmol Vis Sci. 2016 Jul 1;57(9):OCT37-50. doi: 10.1167/iovs.16-19277. PMID 27409495
- [Background] Carrasco-Zevallos OM, Viehland C, Keller B, Draelos M, Kuo AN, Toth CA, Izatt JA. Review of intraoperative optical coherence tomography: technology and applications [Invited]. Biomed Opt Express. 2017 Feb 21;8(3):1607-1637. doi: 10.1364/BOE.8.001607. eCollection 2017 Mar 1. PMID 28663853
- [Background] Viehland C, Keller B, Carrasco-Zevallos OM, Nankivil D, Shen L, Mangalesh S, Viet du T, Kuo AN, Toth CA, Izatt JA. Enhanced volumetric visualization for real time 4D intraoperative ophthalmic swept-source OCT. Biomed Opt Express. 2016 Apr 12;7(5):1815-29. doi: 10.1364/BOE.7.001815. eCollection 2016 May 1. PMID 27231623
- [Background] Carrasco-Zevallos OM, Keller B, Viehland C, Shen L, Waterman G, Todorich B, Shieh C, Hahn P, Farsiu S, Kuo AN, Toth CA, Izatt JA. Live volumetric (4D) visualization and guidance of in vivo human ophthalmic surgery with intraoperative optical coherence tomography. Sci Rep. 2016 Aug 19;6:31689. doi: 10.1038/srep31689. PMID 27538478
- [Background] Chen X, Viehland C, Carrasco-Zevallos OM, Keller B, Vajzovic L, Izatt JA, Toth CA. Microscope-Integrated Optical Coherence Tomography Angiography in the Operating Room in Young Children With Retinal Vascular Disease. JAMA Ophthalmol. 2017 May 1;135(5):483-486. doi: 10.1001/jamaophthalmol.2017.0422. PMID 28384676
- [Background] Li JD, Viehland C, Dhalla AH, Trout R, Raynor W, Kuo AN, Toth CA, Vajzovic LM, Izatt JA. Visualization of surgical maneuvers using intraoperative real-time volumetric optical coherence tomography. Biomed Opt Express. 2023 Jun 29;14(7):3798-3811. doi: 10.1364/BOE.488967. eCollection 2023 Jul 1. PMID 37497507
- [Background] Trout RM, Viehland C, Li JD, Raynor W, Dhalla AH, Vajzovic L, Kuo AN, Toth CA, Izatt JA. Methods for real-time feature-guided image fusion of intrasurgical volumetric optical coherence tomography with digital microscopy. Biomed Opt Express. 2023 Jun 13;14(7):3308-3326. doi: 10.1364/BOE.488975. eCollection 2023 Jul 1. PMID 37497493
- [Background] Li JD, Raynor W, Dhalla AH, Viehland C, Trout R, Toth CA, Vajzovic LM, Izatt JA. Quantitative measurements of intraocular structures and microinjection bleb volumes using intraoperative optical coherence tomography. Biomed Opt Express. 2022 Dec 19;14(1):352-366. doi: 10.1364/BOE.483278. eCollection 2023 Jan 1. PMID 36698674
- [Background] Toth CA. Optical Coherence Tomography and Eye Care. N Engl J Med. 2023 Oct 19;389(16):1526-1529. doi: 10.1056/NEJMcibr2307733. Epub 2023 Sep 21. No abstract available. PMID 37732605